CLINICAL TRIAL: NCT06315140
Title: Building Food Sovereignty, Sustainability and Better Health in Environmentally-impacted Native Americans
Brief Title: Assessing and Addressing Community Exposures to Environmental Contaminants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 22-00248; 1R01ES033545-01 (NIH); 5R01ES033545-02 (NIH)
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Environmental Exposure
Keywords: Ramapough Nation; metals; food; nutrition
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ramapough Lunaape Nation (Experimental): The tribe will be provided with nutrition-rich foods and recipes for nutritious cooking.
  Interventions: Other: Nutrition

INTERVENTIONS:
Other: Nutrition — The intervention will build on the 11-year Tribal-academic partnership with the Ramapough Nation of northern NJ to advance tradition-centered farming practices and management strategies supporting sustainable food systems to relieve local food insecurity. Working with the Ramapough-leased Munsee Three Sisters Medicinal farm (growing produce/crops on clean soil) will provide the tribe with nutrition-rich foods and recipes for nutritious cooking. The interventions aims to return healthy soil on the farm allowing for healthy plant production.

SUMMARY:
The purpose of this study is to build on our equitable, eight-year Tribal-academic partnership with the Ramapough Nation of northern NJ to advance tradition-centered farming practices and management strategies supporting sustainable food systems to relieve local food insecurity and nutritional deficiency, prevent disease and promote health. Furthermore, assessing the extent of environmental contamination, individual toxicant burdens and micronutrient levels and health disorders in Ramapough Tribal members of both sexes as outlined in the following:

* Collect in-person/online survey information on demographics, health and food intake, nutrition, food security, and psychosocial stressors, and perform core anthropometric measurements (i.e., height, weight, body mass index, body circumference and blood pressure) at enrollment on Tribal members to inform health promotion strategies and community actions.
* Determine individual-level contaminant burdens and micronutrient concentrations (e.g., iron, calcium, folate, vitamins) in urine and blood from surveyed (sub-aim 1a) Ramapough Turtle Clan volunteers.
* Test soil, plants and surface water where Turtle Clan residents live, recreate and attend church in Ringwood, NJ using a community-based, citizen scientist approach.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 18 - 80 years old at the time of enrollment
* Living on the streets of Halifax Road, Orange Turnpike, Ramapo Ave, 1st-7th Streets, Mountain Avenue and Fox Hollow Road in Hillburn, NY; Peter's Mine Road, Canon Mine Road, Pipeline Road, Milligan Drive, Cable House Road and Van Dunk Lane in Ringwood, NJ; Stag Hill Road, and Ramapo Brae Lane in Mahwah, NJ
* Willing and able to provide consent

Exclusion Criteria:

* Pregnant women and individuals under 18 or over 80 years old
* Do not live in the identified streets above and/or have lived there for less than 2 years will be excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals with heavy metal contaminants in home water samples | through study completion, an average 2 years
  Outcome measures will be collected using home water samples.
Proportion of individuals with heavy metal and metalloid contaminations in blood biospecimens | through study completion, an average 2 years
  Outcomes measures will be evaluated using blood samples from the Ramapough Lunaape Tribe.
Proportion of individuals with heavy metal and metalloid contaminations in urine biospecimens | through study completion, an average 2 years
  Outcomes measures will be evaluated using urine samples from the Ramapough Lunaape Tribe.
Proportion of individuals with insufficient blood serum micronutrient levels | through study completion, an average 2 years
  Outcome measures will be evaluated using blood serum from the Ramapough Lunaape tribe.
Proportion of individuals with health disorders | through study completion, an average 2 years
  Health status will be assessed using anthropometric measures including blood pressure, body weight, waist circumference, height and Body Mass Index (BMI).

CONTACTS AND LOCATIONS:
Overall Officials: Judith Zelikoff, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Judith.zelikoff@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Judith.zelikoff@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.